CLINICAL TRIAL: NCT02709733
Title: Virtual Rehabilitation for the Treatment of Motivational Deficits in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, George Foussias, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 033-2015
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
Keywords: Virtual Reality; Negative Symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VR Motivation Training (Experimental): Weekly training sessions with a VR motivation treatment 1 hour per week for 8 weeks.
  Interventions: Behavioral: VR Motivation Training

INTERVENTIONS:
Behavioral: VR Motivation Training — Computerized treatment with a virtual reality-based motivation training program, administered for 1 hour per week for 8 weeks.

SUMMARY:
The loss of motivation has emerged as a critical symptom in schizophrenia that is consistently linked to functional disability for affected individuals. Despite advances in treatment, there have not emerged any effective treatments for this loss of motivation, which ultimately hinders our ability to promote recovery for individuals with schizophrenia. To address this critical unmet therapeutic need, this study aims to investigate a novel computerized motivation rehabilitation program using virtual reality to treat motivation loss in schizophrenia.

DETAILED DESCRIPTION:
Motivational deficits have emerged as a critical determinant of functional disability in schizophrenia (SZ). Despite significant advances in our understanding and treatment of the illness, effective therapeutic strategies for motivational deficits have remained elusive. This has ultimately hindered our ability to promote recovery for individuals with SZ so that they can return to their premorbid level of functioning. An emerging therapeutic approach in SZ has utilized computerized remediation strategies, with recent efforts focused on cognitive deficits. To date, however, such a therapeutic strategy has not been developed for the critical motivational deficits in SZ. In light of the detrimental functional consequences of motivational deficits in SZ, there is a clear need for effective therapeutic strategies for the treatment of these motivational deficits experienced by affected individuals. To address this unmet therapeutic need, this pilot therapeutic trial will investigate the efficacy of a novel virtual reality-based motivation rehabilitation program in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 35 years old;
2. DSM-IV diagnosis of Schizophrenia or Schizoaffective Disorder;
3. Outpatients on a stable dose of antipsychotic and other psychotropic medications for the preceding 4 weeks;
4. Minimum Apathy Evaluation Scale (AES) score of 34.

Exclusion Criteria:

1. Diagnosis of other DSM-IV Axis I disorders;
2. History of active substance abuse or dependence in the past 6 months, with the exception of nicotine;
3. History of neurological disease;
4. History of head trauma with loss of consciousness >30 minutes
5. Presence of significant akathisia (a rating of >2 on the Barnes Akathisia Rating Scale (BARS) Global item); or
6. Presence of significant extrapyramidal symptoms (a rating of >2 on >2 items of the Simpson Angus Rating Scale (SARS))
7. Any MRI contraindications.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Apathy Evaluation Scale (AES) | 9 weeks

SECONDARY OUTCOMES:
Scale for the Assessment of Negative Symptoms (SANS) | 9 weeks
Quality of Life Scale (QLS) | 9 weeks
Scale for the Assessment of Positive Symptoms (SAPS) | 9 weeks
Brief Assessment of Cognition in Schizophrenia (BACS) | 9 weeks
Calgary Depression Scale for Schizophrenia (CDSS) | 9 weeks
Simulator Sickness Questionnaire (SSQ) | 9 weeks
Functional Brain Imaging | 9 weeks
  Change in regional brain activity measured with functional MRI
Structural Brain Imaging | 9 weeks
  Changes in brain structure (e.g., white matter tract integrity) measure with structural MRI

CONTACTS AND LOCATIONS:
Overall Officials: George Foussias, MD PhD FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research